CLINICAL TRIAL: NCT02437097
Title: The Effect of Aerobic Exercise and Gaming on Cognitive Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York Institute of Technology (Other)
Responsible Party: Principal Investigator, Peter Douris, Professor of Physical Therapy, New York Institute of Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: BHS-1115
Record Dates: First submitted 2015-05-05; First posted 2015-05-07 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Cognitive Performance in Healthy Volunteers
MeSH Terms: interventions — Exercise; Exergaming

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Aerobic Exercise (Experimental): Participants will perform 30 minutes of cycling at an intensity of 60 to 70% of maximum heart rate based on 220 - their age. The aerobic exercise will utilize a Monarch 818E Monarch Lower Body Ergometer (Monark Exercise, Stockholm, Sweden). Participant's heart rate will be monitored using Polar heart rate monitor.
  Interventions: Other: Aerobic exercise
- Video Gaming (Experimental): Participants will play Brain Age: Train Your Brain in Minutes a Day! on Nintendo 3DS for 30 minutes in a seated resting position.
  Interventions: Other: Video Gaming
- Aerobic Exercise and Video Gaming (Experimental): Participants will perform 30 minutes of cycling at an intensity of 60 to 70% of maximum heart rate based on 220 minus their age on a Monarch ergometer while playing Brain Age: Train Your Brain in Minutes a Day! on a Nintendo 3DS. Participant's heart rate will be monitored using Polar heart rate.
  Interventions: Other: Aerobic exercise and Video Gaming
- Control (Placebo Comparator): Participants will sit quietly for 30 minutes
  Interventions: Other: Control

INTERVENTIONS:
Other: Aerobic exercise — The research design used will be a randomized control trial using a Latin square in order to randomize the treatment conditions. Subjects will take one of four conditions: 1) Aerobic exercise only 2) Aerobic exercise and Gaming simultaneously 3) Gaming only 4) Sitting quietly. All the conditions will take 30 minutes. The independent variables are the four conditions and the dependent variables are the Stroop test and modified Trails B which measure executive function.
  Arms: Aerobic Exercise
Other: Video Gaming — The research design used will be a randomized control trial using a Latin square in order to randomize the treatment conditions. Subjects will take one of four conditions: 1) Aerobic exercise only 2) Aerobic exercise and Gaming simultaneously 3) Gaming only 4) Sitting quietly. All the conditions will take 30 minutes. The independent variables are the four conditions and the dependent variables are the Stroop test and modified Trails B which measure executive function.
  Arms: Video Gaming
Other: Aerobic exercise and Video Gaming — The research design used will be a randomized control trial using a Latin square in order to randomize the treatment conditions. Subjects will take one of four conditions: 1) Aerobic exercise only 2) Aerobic exercise and Gaming simultaneously 3) Gaming only 4) Sitting quietly. All the conditions will take 30 minutes. The independent variables are the four conditions and the dependent variables are the Stroop test and modified Trails B which measure executive function.
  Arms: Aerobic Exercise and Video Gaming
Other: Control — The research design used will be a randomized control trial using a Latin square in order to randomize the treatment conditions. Subjects will take one of four conditions: 1) Aerobic exercise only 2) Aerobic exercise and Gaming simultaneously 3) Gaming only 4) Sitting quietly. All the conditions will take 30 minutes. The independent variables are the four conditions and the dependent variables are the Stroop test and modified Trails B which measure executive function.
  Arms: Control

SUMMARY:
Many studies have examined the effects of aerobic exercise and playing video games effects on cognitive performance, which results of which have shown to increase cognitive performance. Presently, there is limited research regarding the effects of the combination of gaming and exercise on cognitive performance. The purpose of our study is to investigate the effects of playing video games, aerobic exercise, and a combination of gaming and aerobic exercise on cognitive performance. Forty healthy subjects, males and females (18-30 years old) who perform moderate exercise at least two times a week will comprise our sample. The study will be a randomized clinical trial with four independent variables: playing video games, aerobic exercise, a combination of simultaneous gaming and aerobic exercise and a control condition. Aerobic exercise will be performed at an intensity of 60 to 70% of maximum heart rate on a Monarch Lower Body Ergometer. Brain Age Game: Train Your Brain in Minutes a Day! will be played on Nintendo 3DS. Executive function will be measured using the Stroop test and Trails B pre and posttest. Analysis of variance for Stroop test and Trails B will be used. In the event of significant F statistics, a post hoc test analysis will be used. The investigators hypothesize a combination of aerobic exercise and simultaneous gaming will produce the greatest increase in cognitive performance. Furthermore, these beneficial changes can be utilized in rehabilitation protocols designed to improve cognitive functioning.

DETAILED DESCRIPTION:
This study will include 40 subjects, males and females, aged 18-30 years old. Subjects will consist of trained individuals whom log at least two days/week of moderate exercise. The source of participants will come from New York Institute of Technology community. Participants will be selected according to the inclusion/exclusion criteria.Inclusion Criteria:

1. Age range: 18-30 years
2. Good overall health
3. Exercise at least two days/week

Exclusion Criteria:

1. Any cardiopulmonary conditions including asthma within the last 6 months.
2. Any major musculoskeletal injuries (i.e. torn ligaments, bone fractures, etc.) over the last 6 months.
3. Any other health issues that would interfere with a subject's safety during exercise.
4. Any auditory/vestibular impairments.
5. Uncorrected visual problems.

Dr. Douris will be taking the medical history for each prospective subject in order to evaluate for the presence of any of the exclusion criteria. We will use the Physical Activity Readiness Questionnaire (PAR-Q) and our own medical questionnaire. All volunteers will sign the informed consent before participation in the study.

Each subject will require one hour to be tested and to undertake their specific condition which will be randomly assigned. Upon consent form completion subjects will be instructed on how the Stroop and Trails B tests will be administered. The Stroop tests: the subject will be asked to read words of colors, state the colors of various letters to test processing speed, and state the color of the font of a word when the actual word describes a conflicting color to test response inhibition (executive functioning). The Trails B test: the subject is instructed to connect a set of 25 dots as fast as possible while maintaining accuracy. This test provides information about visual search speed, scanning, speed of processing, mental flexibility, and executive functioning. Both tests take approximately 5 minutes to administer. They have both been utilized extensively in the literature to measure changes in executive function as a result of exercise. The subjects will also familiarize themselves with the Brain Age game at the time of consent. Detailed instructions for each testing day are as followed: Pre and Post testing of the Stroop and Trails B tests will occur after each of the four conditions:1) Aerobic exercise only 2) Aerobic exercise and Gaming simultaneously 3) Gaming only 4) Control condition of sitting quietly for 30 minutes. All testing will take place in the School of Health Professions Research Room, Room 507 of the 500 Building.

Acute Bouts of Aerobic Exercise:Participants will perform 30 minutes of cycling at an intensity of 60 to 70% of maximum heart rate based on 220 - their age. The aerobic exercise will utilize a Monarch 818E Monarch Lower Body Ergometer (Monark Exercise, Stockholm, Sweden). Participant's heart rate will be monitored using Polar heart rate monitor.

Acute Bouts of Video Game:Participants will play Brain Age: Train Your Brain in Minutes a Day! on Nintendo 3DS for 30 minutes in a seated resting position.

Acute Bouts of both Aerobic Exercise and Video Games :Participants will perform 30 minutes of cycling at an intensity of 60 to 70% of maximum heart rate based on 220 minus their age on a Monarch ergometer while playing Brain Age: Train Your Brain in Minutes a Day! on a Nintendo 3DS. Participant's heart rate will be monitored using Polar heart rate.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: 18-30 years
2. Good overall health
3. Exercise at least two days/week

Exclusion Criteria:

1. Any cardiopulmonary conditions including asthma within the last 6 months.
2. Any major musculoskeletal injuries (i.e. torn ligaments, bone fractures, etc.) over the last 6 months.
3. Any other health issues that would interfere with a subject's safety during exercise.
4. Any auditory/vestibular impairments.
5. Uncorrected visual problems.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-06; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
The Stroop test | 10 minutes
  : the subject will be asked to read words of colors, state the colors of various letters to test processing speed, and state the color of the font of a word when the actual word describes a conflicting color to test response inhibition (executive functioning).
The Trails B test | 10 minutes
  : the subject is instructed to connect a set of 25 dots as fast as possible while maintaining accuracy. This test provides information about visual search speed, scanning, speed of processing, mental flexibility, and executive functioning.

CONTACTS AND LOCATIONS:
Locations (1):
- New York Institute of Technology, Old Westbury, New York, United States

REFERENCES:
- [Background] O'Leary KC, Pontifex MB, Scudder MR, Brown ML, Hillman CH. The effects of single bouts of aerobic exercise, exergaming, and videogame play on cognitive control. Clin Neurophysiol. 2011 Aug;122(8):1518-25. doi: 10.1016/j.clinph.2011.01.049. Epub 2011 Feb 24. PMID 21353635
- [Background] Byun K, Hyodo K, Suwabe K, Ochi G, Sakairi Y, Kato M, Dan I, Soya H. Positive effect of acute mild exercise on executive function via arousal-related prefrontal activations: an fNIRS study. Neuroimage. 2014 Sep;98:336-45. doi: 10.1016/j.neuroimage.2014.04.067. Epub 2014 May 2. PMID 24799137
- [Background] Chang YK, Chu CH, Wang CC, Song TF, Wei GX. Effect of acute exercise and cardiovascular fitness on cognitive function: an event-related cortical desynchronization study. Psychophysiology. 2015 Mar;52(3):342-51. doi: 10.1111/psyp.12364. Epub 2014 Oct 13. PMID 25308605
- [Background] Yanagisawa H, Dan I, Tsuzuki D, Kato M, Okamoto M, Kyutoku Y, Soya H. Acute moderate exercise elicits increased dorsolateral prefrontal activation and improves cognitive performance with Stroop test. Neuroimage. 2010 May 1;50(4):1702-10. doi: 10.1016/j.neuroimage.2009.12.023. Epub 2009 Dec 16. PMID 20006719
- [Background] Nouchi R, Taki Y, Takeuchi H, Hashizume H, Nozawa T, Kambara T, Sekiguchi A, Miyauchi CM, Kotozaki Y, Nouchi H, Kawashima R. Brain training game boosts executive functions, working memory and processing speed in the young adults: a randomized controlled trial. PLoS One. 2013;8(2):e55518. doi: 10.1371/journal.pone.0055518. Epub 2013 Feb 6. PMID 23405164